CLINICAL TRIAL: NCT00044746
Title: An Open-label, Randomized Study Comparing the Efficacy and Safety of Piperacillin/Tazobactam and Ampicillin/Sulbactam Administered Intravenously in the Empirical Treatment of Foot Infections in Diabetic Inpatients
Brief Title: Study Evaluating the Safety and Efficacy of Piperacillin/Tazobactam and Ampicillin/Sulbactam in Patients With Diabetic Foot Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: 0910X-100468
Record Dates: First submitted 2002-09-04; First posted 2002-09-06 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes Mellitus; Diabetic Foot
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot | interventions — Piperacillin, Tazobactam Drug Combination

INTERVENTIONS:
Drug: Piperacillin/Tazobactam

SUMMARY:
Phase IV Open-Label Foot Infection Study is being conducted to generate comparative Efficacy and Safety data in Diabetic Inpatients.

ELIGIBILITY:
Inclusion Criteria

* Patients with diabetes mellitus
* Inpatient
* Have 1 or more infected ulcer(s) below the ankle

Exclusion Criteria

* Must not have gangrene or severely impaired arterial supply in your foot
* Must not have a bone infection in the area of your ulcer
* Must not have allergies to penicillins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2000-10; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer